CLINICAL TRIAL: NCT02716883
Title: Early Amniotic Membrane Transplantation in Bacterial Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Farabi Eye Hospital (Other)
Responsible Party: Principal Investigator, mohammad soleimani, Assistant Professor, Farabi Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23345
Record Dates: First submitted 2015-08-13; First posted 2016-03-23 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Keratitis of Both Eyes
Keywords: keratitis; AMT; bacterial keratitis; medication
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non AMT (No Intervention): Freshly prepared fortified eye drops (cefazolin 50 mg/mL and amikacin 14 mg/mL) were applied as starting treatment. In the first 3 days, eye drops are applied round the clock followed by drops every 2 h during waking hours until results of laboratory investigation were available.
  After preparation of the culture results, the antimicrobial treatment was narrowed according to bacterial sensitivity. Also topical betamethasone 0.1% four times a day on a tapering weekly dosage until 3-4 weeks is used for all patients. If the patient underwent any tectonic procedure during the treatment such as keratoplasty, cyanoacrylate glue are documented
- AMT (Active Comparator): This group (case group) received above mentioned routine antibiotic therapy followed by double-layer amniotic membrane transplantation 2-5 days after the start of medications and the second group (control group) only received routine antibacterial therapy.
  The AM was trimmed in two layers to fit the corneal ulcer and was placed with its epithelium (basement membrane) side up, secured with 10/0 nylon sutures, supported by a therapeutic contact lens. If the patient underwent any tectonic procedure during the treatment such as keratoplasty, cyanoacrylate glue are documented.
  Interventions: Procedure: AMT

INTERVENTIONS:
Procedure: AMT — The AM was trimmed in two layers to fit the corneal ulcer and was placed with its epithelium (basement membrane) side up, secured with 10/0 nylon sutures, supported by a therapeutic contact lens. The operated eye was patched for 2 h, and then administration of the medical treatment agents was resumed.
  In patients in the case group AMT was performed during days 2-5 of antibiotic therapy when initial clinical response to the treatment was observed.
  Arms: AMT

SUMMARY:
In this study Investigators are going to do early amniotic membrane transplantation (AMT) for bacterial keratitis.

DETAILED DESCRIPTION:
In this study investigators are going to do amniotic membrane transplantation (AMT), early in the first week for bacterial keratitis. Investigators are comparing this technique with no amniotic membrane transplantation (NAMT) in a clinical trial, Inform consent is going to be taken, then the enrolment population is added in the study. Investigators are going to compare the final scar size, the time to scar formation, perforation rate , early need to penetrating keratoplasty (PKP), risk of vision loss (being no light perception (NLP) between two groups.This trial has been approved by the review board in Tehran University of Medical Sciences.( 487/5671)

ELIGIBILITY:
Inclusion Criteria:

Bacterial keratitis being in the first week of diagnosis medically undergoing treatment

Exclusion Criteria:

thinning limbal extension intraocular extension underlying disease Nocardia keratitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Time to scar formation | It needs at most 3 months
  The time keratitis needs for scar to be formed

IPD SHARING:
Plan to Share IPD: No